CLINICAL TRIAL: NCT02824471
Title: Sickle Cell Disease (SCD) Biochip': Towards a Simple and Reliable Way to Monitor Sickle Cell Disease
Brief Title: Sickle Cell Disease Biofluid Chip Technology (SCD BioChip)
Status: Recruiting | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, AOwusu-Ansah, Physician, University Hospitals Cleveland Medical Center
Other Study IDs: 05-14-07C
Record Dates: First submitted 2015-05-27; First posted 2016-07-06 (Estimated); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Biofluidic Chip Technology
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — This is a non-treatment study. The investigators will utilize the leftover blood or cast-off collected from the same blood that will be drawn during participants standard-of-care outpatient or hospital visit.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Minor SCD Group, Ages 12-17: No Intervention. Use of discarded blood/tissue only
  Interventions: Other: SCD Group
- Adult SCD. Ages 18+: No Intervention. Use of discarded blood/tissue only
  Interventions: Other: SCD Group

INTERVENTIONS:
Other: SCD Group — No Intervention. Use of discard blood/tissue

SUMMARY:
'Sickle-shaped' anemia was first clinically described in the US in 1910, and the mutated heritable sickle hemoglobin molecule was identified in 1949. The pathophysiology of SCD is a consequence of abnormal polymerization of sickle hemoglobin (HbS) and its effects on red cell membrane properties, shape, and density, and subsequent critical changes in inflammatory cell and endothelial cell function. Our goal is to understand the impact of CMA abnormalities in SCD, by interrogating a number of recognized interactions in a range of clinical phenotypes.

To date, correlative studies in SCD, by us and others, have range between clinical reports, based on tests, interventions, and chart review of individuals or groups of individuals and, at the other extreme, identification of functional gene polymorphisms based on population studies. The investigators wish to augment these studies through a systematic examination of cellular membrane properties and activation status. Of hematologic disorders, SCD may be unusually susceptible to such an examination.

DETAILED DESCRIPTION:
Novel biofluidic chip technology can investigate surface characteristics that are typically measured with conventional techniques, such as fluorescent activated cell sorting (FACS), immunohistochemistry, or microscopic imaging methods. In FACS, cells of interest are isolated, extensively processed, incubated with a fluorescent-labeled antibody and sorted by optical recognition. In the proposed SCD biofluidic chip (SCD biochip), the interrogating antibody coats the microchannel surface and captures the cell population(s) of interest, without processing, incubation, or in vitro manipulation. The SCD biochip can also quantitate cellular adherence to experimental biological surfaces that are comprised of subcellular components. The SCD biochip is technically simple and experimentally flexible, whereby the population of interest is retained on the chip and quantitated in situ. The microchip system allows retrieval of viable isolated cells for potential downstream processing, analysis, and in vitro culture.

ELIGIBILITY:
Inclusion Criteria

* Male or female ≥12 years of age at the time of consent (enrollment).
* Documentation Sickle Cell Disease, including HbSS or compound heterozygus HbSC- or HbSβ- thalassemia diagnosis as evidenced by one or more clinical features.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal representative and ability for subject to comply with the requirements of the study.

Exclusion Criteria

* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children (≥12 years old) and adults with SCD, including HbSS or compound heterozygus HbSC- or HbSβ- thalassemia will be offered participation. Control samples (HbAA) may be obtained from healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-10 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-05-31 (Estimated)

PRIMARY OUTCOMES:
Develop an SCD Biochip with which to examine key cellular properties and interactions, including RBC and WBC cellular, adhesive, and inflammatory properties, and circulating endothelial and hematopoietic precursor cell characteristics. | 2 years
  Red and white cell adhesion to biomolecules (e.g. laminin, fibronectin, and selectins) will be measured on a microfluidic device, the SCD Biochip. Adhesion will be measured under normal oxygen and low oxygen conditions. Adhesions will be assessed relative to clinical findings, such as hematology parameters, and evidence for vaso-occlusion, pain, inflammation, and vasculopathy in patients with sickle cell disease.endothelial and hematopoietic precursor cells based on membrane properties and adhesion.

SECONDARY OUTCOMES:
Correlate SCD Biochip function in heterogeneous SCD populations, including HbSS and HbSC at a range of ages, and in those with acute and chronic complications and compared with normal controls. | 2 years
  The investigators will examine and validate clinical correlations with these cellular/membrane properties in larger populations of SCD, across a range of phenotypes, using our simple rapid flexible SCD Biochip platform.

CONTACTS AND LOCATIONS:
Overall Officials: Amma Owusu-Ansah, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herrick JB. Peculiar elongated and sickle-shaped red blood corpuscles in a case of severe anemia. 1910. Yale J Biol Med. 2001 May-Jun;74(3):179-84. No abstract available. PMID 11501714
- [Background] PAULING L, ITANO HA, et al. Sickle cell anemia, a molecular disease. Science. 1949 Apr 29;109(2835):443. No abstract available. PMID 18213804
- [Background] Powars DR, Chan LS, Hiti A, Ramicone E, Johnson C. Outcome of sickle cell anemia: a 4-decade observational study of 1056 patients. Medicine (Baltimore). 2005 Nov;84(6):363-376. doi: 10.1097/01.md.0000189089.45003.52. PMID 16267411
- [Background] Nouraie M, Lee JS, Zhang Y, Kanias T, Zhao X, Xiong Z, Oriss TB, Zeng Q, Kato GJ, Gibbs JS, Hildesheim ME, Sachdev V, Barst RJ, Machado RF, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli E, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Goldsmith JC, Gordeuk VR, Gladwin MT; Walk-PHASST Investigators and Patients. The relationship between the severity of hemolysis, clinical manifestations and risk of death in 415 patients with sickle cell anemia in the US and Europe. Haematologica. 2013 Mar;98(3):464-72. doi: 10.3324/haematol.2012.068965. Epub 2012 Sep 14. PMID 22983573
- [Background] Platt OS, Brambilla DJ, Rosse WF, Milner PF, Castro O, Steinberg MH, Klug PP. Mortality in sickle cell disease. Life expectancy and risk factors for early death. N Engl J Med. 1994 Jun 9;330(23):1639-44. doi: 10.1056/NEJM199406093302303. PMID 7993409
- [Background] Platt OS. Easing the suffering caused by sickle cell disease. N Engl J Med. 1994 Mar 17;330(11):783-4. doi: 10.1056/NEJM199403173301110. No abstract available. PMID 8107746
- [Background] Ohene-Frempong K, Weiner SJ, Sleeper LA, Miller ST, Embury S, Moohr JW, Wethers DL, Pegelow CH, Gill FM. Cerebrovascular accidents in sickle cell disease: rates and risk factors. Blood. 1998 Jan 1;91(1):288-94. PMID 9414296
- [Background] West MS, Wethers D, Smith J, Steinberg M. Laboratory profile of sickle cell disease: a cross-sectional analysis. The Cooperative Study of Sickle Cell Disease. J Clin Epidemiol. 1992 Aug;45(8):893-909. doi: 10.1016/0895-4356(92)90073-v. PMID 1624972
- [Background] Charache S, Terrin ML, Moore RD, Dover GJ, Barton FB, Eckert SV, McMahon RP, Bonds DR. Effect of hydroxyurea on the frequency of painful crises in sickle cell anemia. Investigators of the Multicenter Study of Hydroxyurea in Sickle Cell Anemia. N Engl J Med. 1995 May 18;332(20):1317-22. doi: 10.1056/NEJM199505183322001. PMID 7715639
- [Background] Lettre G, Sankaran VG, Bezerra MA, Araujo AS, Uda M, Sanna S, Cao A, Schlessinger D, Costa FF, Hirschhorn JN, Orkin SH. DNA polymorphisms at the BCL11A, HBS1L-MYB, and beta-globin loci associate with fetal hemoglobin levels and pain crises in sickle cell disease. Proc Natl Acad Sci U S A. 2008 Aug 19;105(33):11869-74. doi: 10.1073/pnas.0804799105. Epub 2008 Jul 30. PMID 18667698
- [Background] Milton JN, Rooks H, Drasar E, McCabe EL, Baldwin CT, Melista E, Gordeuk VR, Nouraie M, Kato GR, Minniti C, Taylor J, Campbell A, Luchtman-Jones L, Rana S, Castro O, Zhang Y, Thein SL, Sebastiani P, Gladwin MT; Walk-PHAAST Investigators; Steinberg MH. Genetic determinants of haemolysis in sickle cell anaemia. Br J Haematol. 2013 Apr;161(2):270-8. doi: 10.1111/bjh.12245. Epub 2013 Feb 14. PMID 23406172
- [Background] Bae HT, Baldwin CT, Sebastiani P, Telen MJ, Ashley-Koch A, Garrett M, Hooper WC, Bean CJ, Debaun MR, Arking DE, Bhatnagar P, Casella JF, Keefer JR, Barron-Casella E, Gordeuk V, Kato GJ, Minniti C, Taylor J, Campbell A, Luchtman-Jones L, Hoppe C, Gladwin MT, Zhang Y, Steinberg MH. Meta-analysis of 2040 sickle cell anemia patients: BCL11A and HBS1L-MYB are the major modifiers of HbF in African Americans. Blood. 2012 Aug 30;120(9):1961-2. doi: 10.1182/blood-2012-06-432849. No abstract available. PMID 22936743
- [Background] Milton JN, Sebastiani P, Solovieff N, Hartley SW, Bhatnagar P, Arking DE, Dworkis DA, Casella JF, Barron-Casella E, Bean CJ, Hooper WC, DeBaun MR, Garrett ME, Soldano K, Telen MJ, Ashley-Koch A, Gladwin MT, Baldwin CT, Steinberg MH, Klings ES. A genome-wide association study of total bilirubin and cholelithiasis risk in sickle cell anemia. PLoS One. 2012;7(4):e34741. doi: 10.1371/journal.pone.0034741. Epub 2012 Apr 27. PMID 22558097
- [Background] Dover GJ, Brusilow S, Samid D. Increased fetal hemoglobin in patients receiving sodium 4-phenylbutyrate. N Engl J Med. 1992 Aug 20;327(8):569-70. doi: 10.1056/NEJM199208203270818. No abstract available. PMID 1378939
- [Background] Hebbel RP, Boogaerts MA, Eaton JW, Steinberg MH. Erythrocyte adherence to endothelium in sickle-cell anemia. A possible determinant of disease severity. N Engl J Med. 1980 May 1;302(18):992-5. doi: 10.1056/NEJM198005013021803. PMID 7366623
- [Background] Hebbel RP, Eaton JW, Steinberg MH, White JG. Erythrocyte/endothelial interactions and the vasocclusive severity of sickle cell disease. Prog Clin Biol Res. 1981;55:145-62. PMID 7291188
- [Background] Barabino GA, McIntire LV, Eskin SG, Sears DA, Udden M. Endothelial cell interactions with sickle cell, sickle trait, mechanically injured, and normal erythrocytes under controlled flow. Blood. 1987 Jul;70(1):152-7. PMID 3593962
- [Background] Barabino GA, McIntire LV, Eskin SG, Sears DA, Udden M. Rheological studies of erythrocyte-endothelial cell interactions in sickle cell disease. Prog Clin Biol Res. 1987;240:113-27. PMID 3615482
- [Background] Setty BN, Kulkarni S, Stuart MJ. Role of erythrocyte phosphatidylserine in sickle red cell-endothelial adhesion. Blood. 2002 Mar 1;99(5):1564-71. doi: 10.1182/blood.v99.5.1564. PMID 11861269
- [Background] Kaul DK, Finnegan E, Barabino GA. Sickle red cell-endothelium interactions. Microcirculation. 2009 Jan;16(1):97-111. doi: 10.1080/10739680802279394. PMID 18720225
- [Background] Frenette PS, Atweh GF. Sickle cell disease: old discoveries, new concepts, and future promise. J Clin Invest. 2007 Apr;117(4):850-8. doi: 10.1172/JCI30920. PMID 17404610
- [Background] Belcher JD, Marker PH, Weber JP, Hebbel RP, Vercellotti GM. Activated monocytes in sickle cell disease: potential role in the activation of vascular endothelium and vaso-occlusion. Blood. 2000 Oct 1;96(7):2451-9. PMID 11001897
- [Background] Natarajan M, Udden MM, McIntire LV. Adhesion of sickle red blood cells and damage to interleukin-1 beta stimulated endothelial cells under flow in vitro. Blood. 1996 Jun 1;87(11):4845-52. PMID 8639858
- [Background] Perelman N, Selvaraj SK, Batra S, Luck LR, Erdreich-Epstein A, Coates TD, Kalra VK, Malik P. Placenta growth factor activates monocytes and correlates with sickle cell disease severity. Blood. 2003 Aug 15;102(4):1506-14. doi: 10.1182/blood-2002-11-3422. Epub 2003 Apr 24. PMID 12714517
- [Background] Zennadi R, Chien A, Xu K, Batchvarova M, Telen MJ. Sickle red cells induce adhesion of lymphocytes and monocytes to endothelium. Blood. 2008 Oct 15;112(8):3474-83. doi: 10.1182/blood-2008-01-134346. Epub 2008 Jul 29. PMID 18664622
- [Background] Stone PC, Stuart J, Nash GB. Effects of density and of dehydration of sickle cells on their adhesion to cultured endothelial cells. Am J Hematol. 1996 Jul;52(3):135-43. doi: 10.1002/(SICI)1096-8652(199607)52:33.0.CO;2-U. PMID 8756077
- [Background] Kaul DK, Nagel RL, Chen D, Tsai HM. Sickle erythrocyte-endothelial interactions in microcirculation: the role of von Willebrand factor and implications for vasoocclusion. Blood. 1993 May 1;81(9):2429-38. PMID 8481522
- [Background] Wick TM, Moake JL, Udden MM, Eskin SG, Sears DA, McIntire LV. Unusually large von Willebrand factor multimers increase adhesion of sickle erythrocytes to human endothelial cells under controlled flow. J Clin Invest. 1987 Sep;80(3):905-10. doi: 10.1172/JCI113151. PMID 3497953
- [Background] Brittain HA, Eckman JR, Swerlick RA, Howard RJ, Wick TM. Thrombospondin from activated platelets promotes sickle erythrocyte adherence to human microvascular endothelium under physiologic flow: a potential role for platelet activation in sickle cell vaso-occlusion. Blood. 1993 Apr 15;81(8):2137-43. PMID 8471771
- [Background] Sugihara K, Sugihara T, Mohandas N, Hebbel RP. Thrombospondin mediates adherence of CD36+ sickle reticulocytes to endothelial cells. Blood. 1992 Nov 15;80(10):2634-42. PMID 1384794
- [Background] Barabino GA, Wise RJ, Woodbury VA, Zhang B, Bridges KA, Hebbel RP, Lawler J, Ewenstein BM. Inhibition of sickle erythrocyte adhesion to immobilized thrombospondin by von Willebrand factor under dynamic flow conditions. Blood. 1997 Apr 1;89(7):2560-7. PMID 9116303
- [Background] Finnegan EM, Turhan A, Golan DE, Barabino GA. Adherent leukocytes capture sickle erythrocytes in an in vitro flow model of vaso-occlusion. Am J Hematol. 2007 Apr;82(4):266-75. doi: 10.1002/ajh.20819. PMID 17094094
- [Background] Turhan A, Weiss LA, Mohandas N, Coller BS, Frenette PS. Primary role for adherent leukocytes in sickle cell vascular occlusion: a new paradigm. Proc Natl Acad Sci U S A. 2002 Mar 5;99(5):3047-51. doi: 10.1073/pnas.052522799. PMID 11880644
- [Background] Hebbel RP, Yamada O, Moldow CF, Jacob HS, White JG, Eaton JW. Abnormal adherence of sickle erythrocytes to cultured vascular endothelium: possible mechanism for microvascular occlusion in sickle cell disease. J Clin Invest. 1980 Jan;65(1):154-60. doi: 10.1172/JCI109646. PMID 7350195
- [Background] Solovey A, Lin Y, Browne P, Choong S, Wayner E, Hebbel RP. Circulating activated endothelial cells in sickle cell anemia. N Engl J Med. 1997 Nov 27;337(22):1584-90. doi: 10.1056/NEJM199711273372203. PMID 9371854
- [Background] Strijbos MH, Landburg PP, Nur E, Teerlink T, Leebeek FW, Rijneveld AW, Biemond BJ, Sleijfer S, Gratama JW, Duits AJ, Schnog JJ; CURAMA study group. Circulating endothelial cells: a potential parameter of organ damage in sickle cell anemia? Blood Cells Mol Dis. 2009 Jul-Aug;43(1):63-7. doi: 10.1016/j.bcmd.2009.02.007. Epub 2009 Apr 7. PMID 19356955
- [Background] Hebbel RP, Boogaerts MA, Koresawa S, Jacob HS, Eaton JW, Steinberg MH. Erytrocyte adherence to endothelium as a determinant of vasocclusive severity in sickle cell disease. Trans Assoc Am Physicians. 1980;93:94-9. No abstract available. PMID 7245585
- [Background] van Beem RT, Nur E, Zwaginga JJ, Landburg PP, van Beers EJ, Duits AJ, Brandjes DP, Lommerse I, de Boer HC, van der Schoot CE, Schnog JJ, Biemond BJ; CURAMA Study Group. Elevated endothelial progenitor cells during painful sickle cell crisis. Exp Hematol. 2009 Sep;37(9):1054-9. doi: 10.1016/j.exphem.2009.06.003. Epub 2009 Jun 17. PMID 19539689
- [Background] Jang JE, Hidalgo A, Frenette PS. Intravenous immunoglobulins modulate neutrophil activation and vascular injury through FcgammaRIII and SHP-1. Circ Res. 2012 Apr 13;110(8):1057-66. doi: 10.1161/CIRCRESAHA.112.266411. Epub 2012 Mar 13. PMID 22415018
- [Background] Gurkan UA, Anand T, Tas H, Elkan D, Akay A, Keles HO, Demirci U. Controlled viable release of selectively captured label-free cells in microchannels. Lab Chip. 2011 Dec 7;11(23):3979-89. doi: 10.1039/c1lc20487d. Epub 2011 Oct 14. PMID 22002065
- [Background] Gurkan UA, Tasoglu S, Kavaz D, Demirel MC, Demirci U. Emerging technologies for assembly of microscale hydrogels. Adv Healthc Mater. 2012 Mar;1(2):149-158. doi: 10.1002/adhm.201200011. PMID 23184717
- [Background] Tasoglu S, Gurkan UA, Wang S, Demirci U. Manipulating biological agents and cells in micro-scale volumes for applications in medicine. Chem Soc Rev. 2013 Jul 7;42(13):5788-808. doi: 10.1039/c3cs60042d. PMID 23575660
- [Background] Moon HS, Kwon K, Kim SI, Han H, Sohn J, Lee S, Jung HI. Continuous separation of breast cancer cells from blood samples using multi-orifice flow fractionation (MOFF) and dielectrophoresis (DEP). Lab Chip. 2011 Mar 21;11(6):1118-25. doi: 10.1039/c0lc00345j. Epub 2011 Feb 7. PMID 21298159
- [Background] Rizvi I, Gurkan UA, Tasoglu S, Alagic N, Celli JP, Mensah LB, Mai Z, Demirci U, Hasan T. Flow induces epithelial-mesenchymal transition, cellular heterogeneity and biomarker modulation in 3D ovarian cancer nodules. Proc Natl Acad Sci U S A. 2013 May 28;110(22):E1974-83. doi: 10.1073/pnas.1216989110. Epub 2013 May 3. PMID 23645635
- [Background] Kim KB, Chun H, Kim HC, Chung TD. Red blood cell quantification microfluidic chip using polyelectrolytic gel electrodes. Electrophoresis. 2009 May;30(9):1464-9. doi: 10.1002/elps.200800448. PMID 19340832
- [Background] Gurkan UA, Tasoglu S, Akkaynak D, Avci O, Unluisler S, Canikyan S, Maccallum N, Demirci U. Smart interface materials integrated with microfluidics for on-demand local capture and release of cells. Adv Healthc Mater. 2012 Sep;1(5):661-8. doi: 10.1002/adhm.201200009. Epub 2012 Jul 9. PMID 23184803
- [Background] Machado RF, Barst RJ, Yovetich NA, Hassell KL, Kato GJ, Gordeuk VR, Gibbs JS, Little JA, Schraufnagel DE, Krishnamurti L, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Onyekwere O, Castro OL, Sachdev V, Waclawiw MA, Woolson R, Goldsmith JC, Gladwin MT; walk-PHaSST Investigators and Patients. Hospitalization for pain in patients with sickle cell disease treated with sildenafil for elevated TRV and low exercise capacity. Blood. 2011 Jul 28;118(4):855-64. doi: 10.1182/blood-2010-09-306167. Epub 2011 Apr 28. PMID 21527519
- [Background] Sachdev V, Kato GJ, Gibbs JS, Barst RJ, Machado RF, Nouraie M, Hassell KL, Little JA, Schraufnagel DE, Krishnamurti L, Novelli EM, Girgis RE, Morris CR, Rosenzweig EB, Badesch DB, Lanzkron S, Castro OL, Taylor JG 6th, Hannoush H, Goldsmith JC, Gladwin MT, Gordeuk VR; Walk-PHASST Investigators. Echocardiographic markers of elevated pulmonary pressure and left ventricular diastolic dysfunction are associated with exercise intolerance in adults and adolescents with homozygous sickle cell anemia in the United States and United Kingdom. Circulation. 2011 Sep 27;124(13):1452-60. doi: 10.1161/CIRCULATIONAHA.111.032920. Epub 2011 Sep 6. PMID 21900080
- [Background] Ayyappan, S., et al., Renal Disease in Sickle Cell: Clinically Varied and Associated with Increased Mortality, in American Society of Hematology 2012: Atlanta Georgia
- [Background] Zhang X, Khimji I, Gurkan UA, Safaee H, Catalano PN, Keles HO, Kayaalp E, Demirci U. Lensless imaging for simultaneous microfluidic sperm monitoring and sorting. Lab Chip. 2011 Aug 7;11(15):2535-40. doi: 10.1039/c1lc20236g. Epub 2011 Jun 16. PMID 21677993
- [Background] Zhu X, Zhou N, Zhu J, Zhang Z, Zhang W, Cheng Z, Tu Y, Zhu X. A high-efficiency strategy for synthesizing cyclic polymers of methacryates in one pot. Macromol Rapid Commun. 2013 Jun 25;34(12):1014-9. doi: 10.1002/marc.201300220. Epub 2013 Apr 19. PMID 23606630
- [Background] Yang DH, Yoon GH, Kim SH, Rhee JM, Kim YS, Khang G. Surface and chemical properties of surface-modified UHMWPE powder and mechanical and thermal properties of it impregnated PMMA bone cement, III: effect of various ratios of initiator/inhibitor on the surface modification of UHMWPE powder. J Biomater Sci Polym Ed. 2005;16(9):1121-38. doi: 10.1163/1568562054798572. PMID 16231603
- [Background] Moon S, Ceyhan E, Gurkan UA, Demirci U. Statistical modeling of single target cell encapsulation. PLoS One. 2011;6(7):e21580. doi: 10.1371/journal.pone.0021580. Epub 2011 Jul 21. PMID 21814548
- [Background] Udani M, Zen Q, Cottman M, Leonard N, Jefferson S, Daymont C, Truskey G, Telen MJ. Basal cell adhesion molecule/lutheran protein. The receptor critical for sickle cell adhesion to laminin. J Clin Invest. 1998 Jun 1;101(11):2550-8. doi: 10.1172/JCI1204. PMID 9616226
- [Background] Brown M, Brunson A, Wun T. A method to identify California's sickle-cell disease population and its linkage to the California Cancer Registry. J Registry Manag. 2012 Summer;39(2):53-61. PMID 23599029
- [Background] Luck L, Zeng L, Hiti AL, Weinberg KI, Malik P. Human CD34(+) and CD34(+)CD38(-) hematopoietic progenitors in sickle cell disease differ phenotypically and functionally from normal and suggest distinct subpopulations that generate F cells. Exp Hematol. 2004 May;32(5):483-93. doi: 10.1016/j.exphem.2004.02.003. PMID 15145217
- [Background] Ozdogu H, Sozer O, Boga C, Kozanoglu L, Maytalman E, Guzey M. Flow cytometric evaluation of circulating endothelial cells: a new protocol for identifying endothelial cells at several stages of differentiation. Am J Hematol. 2007 Aug;82(8):706-11. doi: 10.1002/ajh.20904. PMID 17506068
- [Background] Telen MJ. Red blood cell surface adhesion molecules: their possible roles in normal human physiology and disease. Semin Hematol. 2000 Apr;37(2):130-42. doi: 10.1016/s0037-1963(00)90038-6. PMID 10791882
- [Background] Parsons SF, Spring FA, Chasis JA, Anstee DJ. Erythroid cell adhesion molecules Lutheran and LW in health and disease. Baillieres Best Pract Res Clin Haematol. 1999 Dec;12(4):729-45. doi: 10.1053/beha.1999.0050. PMID 10895261
- [Background] El Nemer W, Gauthier E, Wautier MP, Rahuel C, Gane P, Galacteros F, Wautier JL, Cartron JP, Colin Y, Le Van Kim C. Role of Lu/BCAM in abnormal adhesion of sickle red blood cells to vascular endothelium. Transfus Clin Biol. 2008 Feb-Mar;15(1-2):29-33. doi: 10.1016/j.tracli.2008.05.002. Epub 2008 Jun 2. PMID 18514010
- [Background] Chaar V, Picot J, Renaud O, Bartolucci P, Nzouakou R, Bachir D, Galacteros F, Colin Y, Le Van Kim C, El Nemer W. Aggregation of mononuclear and red blood cells through an alpha4beta1-Lu/basal cell adhesion molecule interaction in sickle cell disease. Haematologica. 2010 Nov;95(11):1841-8. doi: 10.3324/haematol.2010.026294. Epub 2010 Jun 18. PMID 20562314
- [Background] Gauthier E, Rahuel C, Wautier MP, El Nemer W, Gane P, Wautier JL, Cartron JP, Colin Y, Le Van Kim C. Protein kinase A-dependent phosphorylation of Lutheran/basal cell adhesion molecule glycoprotein regulates cell adhesion to laminin alpha5. J Biol Chem. 2005 Aug 26;280(34):30055-62. doi: 10.1074/jbc.M503293200. Epub 2005 Jun 23. PMID 15975931
- [Background] Bartolucci P, Chaar V, Picot J, Bachir D, Habibi A, Fauroux C, Galacteros F, Colin Y, Le Van Kim C, El Nemer W. Decreased sickle red blood cell adhesion to laminin by hydroxyurea is associated with inhibition of Lu/BCAM protein phosphorylation. Blood. 2010 Sep 23;116(12):2152-9. doi: 10.1182/blood-2009-12-257444. Epub 2010 Jun 21. PMID 20566895
- [Background] Hillery CA, Du MC, Montgomery RR, Scott JP. Increased adhesion of erythrocytes to components of the extracellular matrix: isolation and characterization of a red blood cell lipid that binds thrombospondin and laminin. Blood. 1996 Jun 1;87(11):4879-86. PMID 8639862
- [Background] De Castro LM, Zennadi R, Jonassaint JC, Batchvarova M, Telen MJ. Effect of propranolol as antiadhesive therapy in sickle cell disease. Clin Transl Sci. 2012 Dec;5(6):437-44. doi: 10.1111/cts.12005. Epub 2012 Oct 17. PMID 23253664
- [Background] Kinney TR, Sleeper LA, Wang WC, Zimmerman RA, Pegelow CH, Ohene-Frempong K, Wethers DL, Bello JA, Vichinsky EP, Moser FG, Gallagher DM, DeBaun MR, Platt OS, Miller ST. Silent cerebral infarcts in sickle cell anemia: a risk factor analysis. The Cooperative Study of Sickle Cell Disease. Pediatrics. 1999 Mar;103(3):640-5. doi: 10.1542/peds.103.3.640. PMID 10049969
- [Background] Stuart MJ, Nagel RL. Sickle-cell disease. Lancet. 2004 Oct 9-15;364(9442):1343-60. doi: 10.1016/S0140-6736(04)17192-4. PMID 15474138
- [Background] Frenette PS. Sickle cell vasoocclusion: heterotypic, multicellular aggregations driven by leukocyte adhesion. Microcirculation. 2004 Mar;11(2):167-77. PMID 15280090
- [Background] Frenette PS. Sickle cell vaso-occlusion: multistep and multicellular paradigm. Curr Opin Hematol. 2002 Mar;9(2):101-6. doi: 10.1097/00062752-200203000-00003. PMID 11844991
- [Background] Chang J, Patton JT, Sarkar A, Ernst B, Magnani JL, Frenette PS. GMI-1070, a novel pan-selectin antagonist, reverses acute vascular occlusions in sickle cell mice. Blood. 2010 Sep 9;116(10):1779-86. doi: 10.1182/blood-2009-12-260513. Epub 2010 May 27. PMID 20508165
- [Background] Wun T, Cordoba M, Rangaswami A, Cheung AW, Paglieroni T. Activated monocytes and platelet-monocyte aggregates in patients with sickle cell disease. Clin Lab Haematol. 2002 Apr;24(2):81-8. doi: 10.1046/j.1365-2257.2002.00433.x. PMID 11985552
- [Background] Cheung AT, Miller JW, Miguelino MG, To WJ, Li J, Lin X, Chen PC, Samarron SL, Wun T, Zwerdling T, Green R. Exchange transfusion therapy and its effects on real-time microcirculation in pediatric sickle cell anemia patients: an intravital microscopy study. J Pediatr Hematol Oncol. 2012 Apr;34(3):169-74. doi: 10.1097/MPH.0b013e31823c27ef. PMID 22278200
- [Background] Wun T, Soulieres D, Frelinger AL, Krishnamurti L, Novelli EM, Kutlar A, Ataga KI, Knupp CL, McMahon LE, Strouse JJ, Zhou C, Heath LE, Nwachuku CE, Jakubowski JA, Riesmeyer JS, Winters KJ. A double-blind, randomized, multicenter phase 2 study of prasugrel versus placebo in adult patients with sickle cell disease. J Hematol Oncol. 2013 Feb 17;6:17. doi: 10.1186/1756-8722-6-17. PMID 23414938
- [Background] Wood KC, Hebbel RP, Granger DN. Endothelial cell P-selectin mediates a proinflammatory and prothrombogenic phenotype in cerebral venules of sickle cell transgenic mice. Am J Physiol Heart Circ Physiol. 2004 May;286(5):H1608-14. doi: 10.1152/ajpheart.01056.2003. Epub 2004 Jan 2. PMID 14704223
- [Background] Wood K, Russell J, Hebbel RP, Granger DN. Differential expression of E- and P-selectin in the microvasculature of sickle cell transgenic mice. Microcirculation. 2004 Jun;11(4):377-85. doi: 10.1080/10739680490437559. PMID 15280076
- [Background] Hidalgo A, Chang J, Jang JE, Peired AJ, Chiang EY, Frenette PS. Heterotypic interactions enabled by polarized neutrophil microdomains mediate thromboinflammatory injury. Nat Med. 2009 Apr;15(4):384-91. doi: 10.1038/nm.1939. Epub 2009 Mar 22. PMID 19305412
- [Background] Canalli AA, Proenca RF, Franco-Penteado CF, Traina F, Sakamoto TM, Saad ST, Conran N, Costa FF. Participation of Mac-1, LFA-1 and VLA-4 integrins in the in vitro adhesion of sickle cell disease neutrophils to endothelial layers, and reversal of adhesion by simvastatin. Haematologica. 2011 Apr;96(4):526-33. doi: 10.3324/haematol.2010.032912. Epub 2010 Dec 20. PMID 21173096
- [Background] Almeida CB, Scheiermann C, Jang JE, Prophete C, Costa FF, Conran N, Frenette PS. Hydroxyurea and a cGMP-amplifying agent have immediate benefits on acute vaso-occlusive events in sickle cell disease mice. Blood. 2012 Oct 4;120(14):2879-88. doi: 10.1182/blood-2012-02-409524. Epub 2012 Jul 25. PMID 22833547
- [Background] Matsui NM, Borsig L, Rosen SD, Yaghmai M, Varki A, Embury SH. P-selectin mediates the adhesion of sickle erythrocytes to the endothelium. Blood. 2001 Sep 15;98(6):1955-62. doi: 10.1182/blood.v98.6.1955. PMID 11535535
- [Background] Enenstein J, Milbauer L, Domingo E, Wells A, Roney M, Kiley J, Wei P, Hebbel RP. Proinflammatory phenotype with imbalance of KLF2 and RelA: risk of childhood stroke with sickle cell anemia. Am J Hematol. 2010 Jan;85(1):18-23. doi: 10.1002/ajh.21558. PMID 19957349
- [Background] Kato GJ, Hebbel RP, Steinberg MH, Gladwin MT. Vasculopathy in sickle cell disease: Biology, pathophysiology, genetics, translational medicine, and new research directions. Am J Hematol. 2009 Sep;84(9):618-25. doi: 10.1002/ajh.21475. PMID 19610078
- [Background] Safaya S, Steinberg MH, Klings ES. Monocytes from sickle cell disease patients induce differential pulmonary endothelial gene expression via activation of NF-kappaB signaling pathway. Mol Immunol. 2012 Feb;50(1-2):117-23. doi: 10.1016/j.molimm.2011.12.012. Epub 2012 Jan 20. PMID 22264835
- [Background] Shiu YT, Udden MM, McIntire LV. Perfusion with sickle erythrocytes up-regulates ICAM-1 and VCAM-1 gene expression in cultured human endothelial cells. Blood. 2000 May 15;95(10):3232-41. PMID 10807794
- [Background] Sowemimo-Coker SO, Meiselman HJ, Francis RB Jr. Increased circulating endothelial cells in sickle cell crisis. Am J Hematol. 1989 Aug;31(4):263-5. doi: 10.1002/ajh.2830310409. PMID 2741925
- [Background] Solovey A, Gui L, Ramakrishnan S, Steinberg MH, Hebbel RP. Sickle cell anemia as a possible state of enhanced anti-apoptotic tone: survival effect of vascular endothelial growth factor on circulating and unanchored endothelial cells. Blood. 1999 Jun 1;93(11):3824-30. PMID 10339489
- [Background] Anjum F, Lazar J, Zein J, Jamaleddine G, Demetis S, Wadgaonkar R. Characterization of altered patterns of endothelial progenitor cells in sickle cell disease related pulmonary arterial hypertension. Pulm Circ. 2012 Jan-Mar;2(1):54-60. doi: 10.4103/2045-8932.94834. PMID 22558520
- [Background] Boga C, Kozanoglu I, Ozdogu H, Sozer O, Sezgin N, Bakar C. Alterations of circulating endothelial cells after apheresis in patients with sickle cell disease: a potential clue for restoration of pathophysiology. Transfus Apher Sci. 2010 Dec;43(3):273-279. doi: 10.1016/j.transci.2010.09.015. Epub 2010 Oct 15. PMID 20951649
- [Background] Samsel L, Dagur PK, Raghavachari N, Seamon C, Kato GJ, McCoy JP Jr. Imaging flow cytometry for morphologic and phenotypic characterization of rare circulating endothelial cells. Cytometry B Clin Cytom. 2013 Nov-Dec;84(6):379-89. doi: 10.1002/cyto.b.21088. Epub 2013 Mar 29. PMID 23554273
- [Background] Nayak L, Goduni L, Takami Y, Sharma N, Kapil P, Jain MK, Mahabeleshwar GH. Kruppel-like factor 2 is a transcriptional regulator of chronic and acute inflammation. Am J Pathol. 2013 May;182(5):1696-704. doi: 10.1016/j.ajpath.2013.01.029. Epub 2013 Mar 13. PMID 23499374
- [Background] Lin Z, Natesan V, Shi H, Dong F, Kawanami D, Mahabeleshwar GH, Atkins GB, Nayak L, Cui Y, Finigan JH, Jain MK. Kruppel-like factor 2 regulates endothelial barrier function. Arterioscler Thromb Vasc Biol. 2010 Oct;30(10):1952-9. doi: 10.1161/ATVBAHA.110.211474. Epub 2010 Jul 22. PMID 20651277
- [Background] Mahabeleshwar GH, Qureshi MA, Takami Y, Sharma N, Lingrel JB, Jain MK. A myeloid hypoxia-inducible factor 1alpha-Kruppel-like factor 2 pathway regulates gram-positive endotoxin-mediated sepsis. J Biol Chem. 2012 Jan 6;287(2):1448-57. doi: 10.1074/jbc.M111.312702. Epub 2011 Nov 22. PMID 22110137
- [Background] Paulson RF, Shi L, Wu DC. Stress erythropoiesis: new signals and new stress progenitor cells. Curr Opin Hematol. 2011 May;18(3):139-45. doi: 10.1097/MOH.0b013e32834521c8. PMID 21372709
- [Background] Connes P, Coates TD. Autonomic nervous system dysfunction: implication in sickle cell disease. C R Biol. 2013 Mar;336(3):142-7. doi: 10.1016/j.crvi.2012.09.003. Epub 2012 Oct 16. PMID 23643396
- [Background] Sangkatumvong S, Khoo MC, Coates TD. Abnormal cardiac autonomic control in sickle cell disease following transient hypoxia. Annu Int Conf IEEE Eng Med Biol Soc. 2008;2008:1996-9. doi: 10.1109/IEMBS.2008.4649581. PMID 19163084
- [Background] Lucas D, Bruns I, Battista M, Mendez-Ferrer S, Magnon C, Kunisaki Y, Frenette PS. Norepinephrine reuptake inhibition promotes mobilization in mice: potential impact to rescue low stem cell yields. Blood. 2012 Apr 26;119(17):3962-5. doi: 10.1182/blood-2011-07-367102. Epub 2012 Mar 14. PMID 22422821
- [Background] de Jong K, Emerson RK, Butler J, Bastacky J, Mohandas N, Kuypers FA. Short survival of phosphatidylserine-exposing red blood cells in murine sickle cell anemia. Blood. 2001 Sep 1;98(5):1577-84. doi: 10.1182/blood.v98.5.1577. PMID 11520810
- [Background] de Jong K, Larkin SK, Styles LA, Bookchin RM, Kuypers FA. Characterization of the phosphatidylserine-exposing subpopulation of sickle cells. Blood. 2001 Aug 1;98(3):860-7. doi: 10.1182/blood.v98.3.860. PMID 11468189
- [Background] Manodori AB, Barabino GA, Lubin BH, Kuypers FA. Adherence of phosphatidylserine-exposing erythrocytes to endothelial matrix thrombospondin. Blood. 2000 Feb 15;95(4):1293-300. PMID 10666202
- [Background] Kuypers FA, Lewis RA, Hua M, Schott MA, Discher D, Ernst JD, Lubin BH. Detection of altered membrane phospholipid asymmetry in subpopulations of human red blood cells using fluorescently labeled annexin V. Blood. 1996 Feb 1;87(3):1179-87. PMID 8562945
- [Background] Schwartz RS, Tanaka Y, Fidler IJ, Chiu DT, Lubin B, Schroit AJ. Increased adherence of sickled and phosphatidylserine-enriched human erythrocytes to cultured human peripheral blood monocytes. J Clin Invest. 1985 Jun;75(6):1965-72. doi: 10.1172/JCI111913. PMID 4008648
- [Background] Setty BN, Kulkarni S, Dampier CD, Stuart MJ. Fetal hemoglobin in sickle cell anemia: relationship to erythrocyte adhesion markers and adhesion. Blood. 2001 May 1;97(9):2568-73. doi: 10.1182/blood.v97.9.2568. PMID 11313243